CLINICAL TRIAL: NCT03027349
Title: Serum Calcium to Phosphorous Ratio (Ca/P) as a Simple, Inexpensive Screening Tool in the Diagnosis of Primary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Manuela Simoni, Director, Azienda USL Modena
Other Study IDs: Primary hyperparathyroidism
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: Patients aged between 18-90 years old with primary hyperparathyroidism who had been diagnosed in the Unit of Endocrinology of the University of Modena and Reggio Emilia.
  The exclusion criteria will be:
  * age younger than 18 years
  * renal and liver failure and insufficiency
  * active metabolic bone disease (such as Paget's disease of the bone, osteomalacia, rickets, etc)
  * any type of cancer
  * malnutrition, severe obesity (BMI > 40 kg/m2) and malabsorption
  * transplantation
  * sarcoidosis
  * endocrinological disorders such as hypercortisolism, diabetes insipidus, hyperthyroidism, pseudohypoparathyroidism
  * familial hypocalciuric hypercalcemia
  * hypophosphoremia sustained by genetic causes or secondary to other causes.
  Interventions: Other: No intervention are provided
- Control group: Patients that underwent biochemical examination by primary care physician or by endocrinologist in order to assess their parathyroid function and calcium metabolism state with results into the normal ranges.
  The exclusion criteria will be:
  * age younger than 18 years
  * renal and liver failure and insufficiency
  * active metabolic bone disease (such as Paget's disease of the bone, osteomalacia, rickets, etc)
  * any type of cancer
  * malnutrition, severe obesity (BMI > 40 kg/m2) and malabsorption
  * transplantation
  * sarcoidosis
  * endocrinological disorders such as hypercortisolism, diabetes insipidus, hyperthyroidism, pseudohypoparathyroidism
  * familial hypocalciuric hypercalcemia
  * hypophosphoremia sustained by genetic causes or secondary to other causes.
  Interventions: Other: No intervention are provided

INTERVENTIONS:
Other: No intervention are provided

SUMMARY:
Background:

Primary hyperparathyroidism (PHPT) is often overlooked and underdiagnosed. At present the diagnosis of PHPT remains challenging and is based on serum calcium (Ca) and PTH.

As serum Ca and phosphorous (P) are inversely related in PHPT, the Ca/P ratio might be considered a good candidate tool in the diagnosis of PHPT.

AIM: The aim of this study is to investigate the diagnostic value of the Ca/P ratio in the diagnosis of PHPT.

Study design: Retrospective, observational, cross-sectional, case-control clinical trial will be carried out.

Biochemical measurements will include PTH, Vitamin D, serum Ca, P, albumin, and creatinine.

ELIGIBILITY:
Inclusion Criteria:

* elevated parathormone serum levels
* normal or elevated calcium serum levels

Exclusion Criteria:

* age younger than 18 years
* renal and liver failure and insufficiency
* active metabolic bone disease (such as Paget's disease of the bone, osteomalacia, rickets, etc)
* any type of cancer
* malnutrition, severe obesity (BMI > 40 kg/m2) and malabsorption
* transplantation
* sarcoidosis
* endocrinological disorders such as hypercortisolism, diabetes insipidus, hyperthyroidism, pseudohypoparathyroidism
* familial hypocalciuric hypercalcemia
* hypophosphoremia sustained by genetic causes or secondary to other causes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of primary hyperparathyroidism
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2011-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Calcium | Enrollment time
  Assay performed at the moment of diagnosis

SECONDARY OUTCOMES:
Phosphorus | Enrollment time
  Assay performed at the moment of diagnosis
Parathormone | Enrollment time
  Assay performed at the moment of diagnosis
Creatinine | Enrollment time
  Assay performed at the moment of diagnosis
Albumine | Enrollment time
  Assay performed at the moment of diagnosis
Vitamin D | Enrollment time
  Assay performed at the moment of diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL of Modena, Modena, Modena, Italy